CLINICAL TRIAL: NCT06534710
Title: Ffect of Electronic Moxibustion Apparatus on Pain Degree and Wound Healing of Patients After Craniocerebral Surgery
Brief Title: Effect of Electronic Moxibustion Apparatus on Pain Degree and Wound Healing of Patients After Craniocerebral Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KY-2024-117
Record Dates: First submitted 2024-06-30; First posted 2024-08-02 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Patients Undergoing Craniocerebral Surgery
Keywords: Craniocerebral surgery; Electronic moxibustion; Wound healing;; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Creditease Medical Device Technology，YXB-AJY-06
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): On the basis of the control group, an electronic moxibustion instrument was used every day (CreditEase Medical Device Technology, YXB-AJY-06) : The patient was placed in a comfortable lying position and the surgical incision area was fully exposed. The nurse placed the moxibustion tablets on the moxibustion head of the electronic moxibustion instrument, and the moxibustion head was connected to the electronic moxibustion treatment instrument through a wire. The moxibustion temperature should be slightly red on the skin and the patient should tolerate it. The total intervention time was 5 days, and the relevant study data at discharge were recorded if the patient was discharged early
  Interventions: Device: electronic moxibustion apparatus
- control group (No Intervention): The routine nursing plan was adopted. (1) Pain knowledge education, including understanding of pain and analgesic drugs, pain assessment methods, selection of analgesic drugs, etc. within 24 hours of admission and before and after surgery, to alleviate patients' fear and anxiety about pain; ② After surgery, choose the appropriate position, gently turn over, and try to avoid pain caused by the change of position and pressure on the affected side; ③ After the gauze or dressing was removed from the surgical incision, the nurse disinfected the surgical incision twice a day with iodophor cotton swabs, observed the healing of the wound at the surgical incision every day, and reported to the doctor in time if there was blood or fluid leakage.

INTERVENTIONS:
Device: electronic moxibustion apparatus — The experimental group used the electronic moxibustion instrument every day on the basis of the control group
  Arms: experimental group

SUMMARY:
According to statistics, about 70% to 84% of patients after craniocerebral surgery will have moderate to severe wound pain, especially within 24h after surgery [1]. Pain can reduce the comfort of patients, affect the speed of incision healing, and interfere with the prognosis and rehabilitation effect in the later stage. At present, non-steroidal drugs are often used clinically for analgesic intervention, but the use of drugs often brings gastrointestinal discomfort such as nausea and vomiting, and is easy to produce dependence. In addition, redness, swelling, fluid leakage, cracking or no hair growth around the incision are prone to poor surgical incision healing after cranial surgery [2]. Poor healing of surgical incision will not only lead to prolonged hospital stay, increase hospital costs, but also bring trauma and pain to patients, and even induce medical disputes. Moxibustion is an important branch of TCM physiotherapy. It has the functions of warming, clearing and dispersing. It can inhibit inflammation through various ways, relieve local pain and edema, and its effect is mild. At present, moxibustion is mostly used to promote the recovery of urinary or gastrointestinal functions, and the healing of surgical wounds after anal fistula or perianal abscess. There are no relevant studies on its application to surgical incision in patients after craniocerebral surgery. The effect of moxibustion on improving the pain and healing of surgical incision in patients after craniocerebral surgery is still unknown. Considering the disadvantages of traditional moxibustion, such as inconvenient operation, easy burn at high temperature and environmental pollution by moxibustion smoke, this study will use an electronic moxibustion instrument. Patients on the third day after craniectomy were divided into two groups by random number table method. Patients in the control group were given routine care; patients in the experimental group were irradiated with the postoperative incision with an electronic moxibustion instrument every day on the basis of the control group. The pain score at the surgical incision, the healing score value of the surgical incision, the healing time of the incision and the occurrence of adverse events during the incision healing were compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients on the third day after craniocerebral surgery; ② Patients with vital signs and stable condition for more than 24 hours; (3) Meet the requirements of medical research ethics, and the subjects voluntarily join the clinical study and sign the informed consent; (4) The expected duration of hospitalization is > 3 days; ⑤ Age > 18 years old;

Exclusion Criteria:

① Patients with serious heart, lung, liver, kidney and other vital organ dysfunction; ② Female patients in lactation period, menstrual period, pregnancy period or allergic constitution; Exclusion criteria: ① Patients or their family members should be excluded from this study in time due to disputes with the hospital during diagnosis or treatment (including requests for early transfer and termination of treatment).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
pain score | Baseline and 5 days after intervention
  Awake patients were scored with numeric rating scales (NRS). 0 was classified as no pain, 1-3 was classified as mild pain (pain did not affect sleep), 4-6 was classified as moderate pain (pain did not affect sleep), and 7-10 was classified as severe pain (unable to fall asleep or wake up with pain). Patients with coma or disturbance of consciousness were treated with behavioral pain scale (specific score).

SECONDARY OUTCOMES:
Incision healing score | Baseline and 5 days after intervention
  Scalp incision healing criteria were evaluated, with a score of 3 to 13,3 to 5 as incision healing, and ≥6 as poor incision healing. The surgical incisions were evaluated and recorded by nurses daily according to the wound healing scale.
Incision healing time | 4 weeks after intervention
  According to the scalp incision healing standard, when the score is less than 6 points, it is considered as surgical incision healing. If the surgical incision had not healed at the time of discharge, the wound healing score at discharge was recorded.
The occurrence of adverse events in incision healing | Baseline and 5 days after intervention
  Adverse reactions related to surgical incision healing (such as suppuration, crusts, tension blisters, skin ecchymosis around the incision or incision split, etc.), severity and treatment methods were included in the study during the study process, and their safety was objectively evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- the Fourth Affiliated Hospital of School of Medicine, and International School of Medicine, International Institutes of Medicine，Zhejiang University, Yiwu, Zhejiang, China